CLINICAL TRIAL: NCT02567331
Title: An Open-label Study of the Safety, Tolerability, and Response Rate of Xeloda in Treatment-naïve Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Capecitabine (Xeloda) in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18017
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

ARMS (1):
- Capecitabine (Experimental): Participants will receive oral capecitabine 1250 milligrams per square meter (mg/m^2) twice daily for 14 days followed by 7 day rest period for 6 cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Participants will receive 1250 mg/m^2 capecitabine administered twice daily as oral tablets for 14 days followed by a 7 day rest period for up to 6 treatment cycles.
  Other Names: Xeloda

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacoeconomics of oral capecitabine in patients with metastatic colorectal cancer. The anticipated time on study treatment is 3-12 months, and the target sample size is 28 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to (>=) 18 years of age
* Metastatic colorectal cancer

Exclusion Criteria:

* Previous cytotoxic chemotherapy or immunotherapy for advanced or metastatic disease
* Central nervous system and bone metastases
* Moderate or severe renal impairment
* Clinically significant cardiac disease
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication
* Malignancy within the last 5 years, except cured basal cell cancer of skin and cured cancer in situ of uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to approximately 1.5 years
Response rate, ie, percentage of participants with complete, partial, and overall response | up to approximately 1.5 years

SECONDARY OUTCOMES:
Pharmacoeconomic analysis: Treatment-related and AE-related spending/savings\n | up to approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Stara Zagora